CLINICAL TRIAL: NCT00327652
Title: Phase 1 Dose-Escalation Study of Safety and Tolerability of Intravenous CRS-100 in Adults With Carcinoma and Liver Metastases
Brief Title: Study of Safety and Tolerability of Intravenous CRS-100 in Adults With Carcinoma and Liver Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anza Therapeutics, Inc. (Industry)
Responsible Party: David N. Cook, PhD, Anza Therapeutics, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAC05001
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2008-04

CONDITIONS: Neoplasm Metastasis; Liver Neoplasms; Carcinoma
Keywords: carcinoma; liver; hepatic; metastasis; Listeria
MeSH Terms: conditions — Neoplasm Metastasis; Liver Neoplasms; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CRS-100 — Live-attenuated Listeria monocytogenes

SUMMARY:
This clinical trial evaluated the safety and tolerability of CRS-100, an investigational agent containing a live-attenuated strain of Listeria monocytogenes (Lm). CRS-100 is attenuated by genetic modification to limit cell to cell spread and invasion of liver cells. These attenuations result in decreased virulence of CRS-100 in mice but retain the ability of the investigational agent to stimulate immunity in test animals and generate anti-tumor activity in mice. The primary objective of this study was to determine the maximum tolerated dose (MTD) and to explore the safety profile of a single intravenous dose of CRS-100 in consenting volunteers. Immunological response to CRS-100 and tumor status of study participants were also measured. Participation in this first clinical trial with CRS-100 was restricted to adults with carcinoma refractory to standard treatment (or for whom no standard treatment is available) and who additionally had liver metastases.

DETAILED DESCRIPTION:
Patients who consented to participate in the study were evaluated for eligibility according to their medical history, physical examination, blood testing, and computed tomography (CT) scan of thorax, abdomen, and pelvis. Those patients who qualified for the study received a single intravenous dose of CRS-100 on study day 1, after which they remained in the hospital for five days for safety monitoring of health status, including serial blood collections. Study participants returned for out-patient follow-up for further blood tests and additional monitoring of safety and immune response to CRS-100. At day 56, after administration of CRS-100, participants had a repeat CT scan to measure tumor size, and they were then discharged from the study.

ELIGIBILITY:
Inclusion Criteria (abbreviated):

1. Documented carcinoma refractory to standard treatment (or for whom no standard treatment is available). Hepatocellular carcinoma (HCC) is not allowed.
2. Hepatic metastases
3. ECOG Performance Status of 0 or 1, or Karnofsky Performance Status (KPS) of 80% to 100%.
4. Adequate organ function as defined by clinical hematology and chemistry assays.

Exclusion Criteria (abbreviated):

1. Known central nervous system metastases.
2. History of allergic reactions attributed to sulfa or beta-lactam antibiotics.
3. Cardiac conditions associated with high- or moderate-risk of endocarditis.
4. Intra-arterial hepatic catheter, hepatic cirrhosis, or clinically relevant ascites.
5. Artificial (prosthetic) joint or other artificial implant or devices that cannot easily be removed.
6. Known coagulation disorder or recent thromboembolic event.
7. Use of immunosuppressive agent, chemotherapy, or radiation therapy within 28 days prior to CRS-100; bone marrow or stem cell transplant or a major organ allograft; autoimmune disease.
8. Current history of gallstones or kidney stones.
9. Infection with HIV, human t-lymphotropic virus type 1 (HTLV-1), hepatitis c virus (HCV), or hepatitis b virus (HBV).
10. Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-10; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) for 7 days after dosing | 7 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Mary Crowley Medical Research Center, Dallas, Texas